CLINICAL TRIAL: NCT01008813
Title: A Randomized Phase II Trial to Evaluate the Immunogenicity and Safety of an Adjuvanted A(H1N1)v Influenza Vaccine and a Non-adjuvanted A(H1N1)v Influenza Vaccine in HIV-infected Patients (ANRS 151 Hifluvac)
Brief Title: Clinical Trial to Evaluate the Immunogenicity and Safety of an Adjuvanted A(H1N1)v Influenza Vaccine and a Non-adjuvanted A(H1N1)v Influenza Vaccine in HIV-infected Patients (ANRS 151 Hifluvac)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-016226-13
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections
Keywords: HIV infection; adjuvanted and non-adjuvanted A(H1N1)v influenza vaccine; immunogenicity; safety
MeSH Terms: conditions — HIV Infections | interventions — pandemrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adjuvanted A(H1N1)v influenza vaccine (Experimental): Two injections at day 0 and day 21
  Interventions: Biological: adjuvanted A(H1N1)v influenza vaccine
- non-adjuvanted A(H1N1)v influenza vaccine (Experimental): Two injection at day 0 and day 21
  Interventions: Biological: non-adjuvanted A(H1N1)v influenza vaccine

INTERVENTIONS:
Biological: adjuvanted A(H1N1)v influenza vaccine — Two intramuscular injections at day 0 and day 21 of FLU D-PAN H1N1 [A/California/7/2009 (H1N1)v] (3,8 microgram) adjuvanted with AS 03A
  Other Names: Pandemrix
  Arms: adjuvanted A(H1N1)v influenza vaccine
Biological: non-adjuvanted A(H1N1)v influenza vaccine — Two intramuscular injections at day 0 and day 21 of FLU D-PAN H1N1 [A/California/7/2009 (H1N1)v] (15 microgram)
  Arms: non-adjuvanted A(H1N1)v influenza vaccine

SUMMARY:
A 1-year multicenter, randomized, single-blinded, phase II trial, stratified on HAART. The purpose of this trial is to evaluate the immunogenicity and safety of a A(H1N1)French National Agency for Research on AIDS and Viral Hepatitis influenza vaccine, administered with or without adjuvant, in HIV-infected patients after one or two injections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to give written consent
* Covered by French Social Security
* HIV-infected (infection attested by the patient's chart)
* Patients treated by HAART for at least 6 months, with a viral load inferior to 50 copies/mL on at least 2 last visits
* Patients without any treatment for HIV for at least 6 months and without any indication to start a treatment in the following 3 months
* Patients followed for their HIV-infection in an ANRS center and whose home is close to the center in case of influenza-like illness, consultation and hospitalization in the center where he is followed if necessary
* For women with childbearing potential, using an effective method of contraception, and willing to undergo urine pregnancy tests prior to each vaccination.

Exclusion Criteria:

* Pregnancy
* Receipt of chemotherapy, immunotherapy (IL2, IL7, IV Ig), or corticosteroids within 3 months prior to enrolment
* Thrombopenia inferior to 20 000/mm3
* Febrile episode (at least 38°C rectal or if at least 37,5°C measured orally) within one week prior to vaccination
* Opportunistic infection (treated for less than 1 month)
* Co-infection with HCV and treated with IFNa
* Influenza (clinically or virologically documented) in the last 6 months
* History of documented auto-immune disease (lupus, systemic inflammatory disease, ...)
* Child C cirrhosis
* Solid organ transplant recipient
* Intolerance to 1 component of the vaccine
* Other immunization received within 3 weeks prior to inclusion or planned until after the last vaccine injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity and safety of a A(H1N1)v influenza vaccine, administered with or without adjuvant, in HIV-infected patients after two injections. | Day 42

SECONDARY OUTCOMES:
To evaluate the safety (local and general adverse events) between the two study vaccines | From week 0 to week 48
To evaluate the immunogenicity of a A(H1N1)v influenza vaccine, administered with or without adjuvant, in HIV-infected patients receiving antiretroviral therapy or not | Day 21 and Day 42
To describe the factors influencing the response to the vaccine (such as age, sex, tobacco use, HAART, CD4 count and nadir, HIV viral load, ...) | From week 0 to week 48
To compare the sustainability of the immune response induced by two injections of the study | Day 21 and Day 42
To explore the post-vaccinal cellular immune response of the two study vaccines | Day 42
To compare the consequences of the A(H1N1)v influenza vaccine, with or without adjuvant, on the HIV infection parameters (CD4 count, HIV viral load) | Week 48
To assess vaccination failures and describe the clinical presentation of influenza in the study population | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, Principal Investigator — Centre d'investigation clinique de vaccinologie Cochin-Pasteur, Hôpital Cochin, Paris, France
Locations (6):
- France (6):
  - Hôpital Henri Mondor, Créteil
  - Hopital du Kremlin Bicêtre Service de médecine interne, Kremlin Bicëtre
  - Hôpital Saint-Louis, Paris
  - Service des Maladies Infectieuses et Tropicales, Hopital Tenon, Paris
  - CIC de Vaccinologie Cochin Pasteur, hôpital Cochin, Paris
  - Hôpital Gustave Dron, Service Maladies Infectieuses, Tourcoing

REFERENCES:
- See also: legal sponsor's website — http://www.anrs.fr